CLINICAL TRIAL: NCT00739414
Title: A Phase IA, Dose-escalating Study of LBH589 Administered Intravenously in Adult Patients With Advanced Solid Tumors
Brief Title: Dose-escalating Study of LBH589 in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLBH589A1101
Record Dates: First submitted 2008-08-18; First posted 2008-08-21 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2010-03

CONDITIONS: Cancer; Advanced Solid Tumor
Keywords: Histone Deacetylases; HDAC inhibitor; LBH589; Advanced solid tumor; Adult
MeSH Terms: conditions — Neoplasms | interventions — Panobinostat

ARMS (1):
- LBH589 (Panobinostat) (Experimental)
  Interventions: Drug: LBH589

INTERVENTIONS:
Drug: LBH589 — 10, 15, 20 mg/m2, i.v. on day 1 and 8 of each 21 day cycle
  Other Names: Panobinostat

SUMMARY:
This study will characterize the safety, tolerability, biological activity, and pharmacokinetics of LBH589 in Japanese patients with advanced solid tumors whose disease has progressed despite standard therapies, or for whom no standard therapy exists.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologically or cytologically confirmed, advanced solid tumors whose disease has progressed despite available standard therapies, or for which no standard therapy exists.
2. At least one measurable or non-measurable lesion as defined by modified RECIST Criteria for solid tumors
3. Age ≥20 years old
4. World Health Organization (WHO) Performance Status of ≤2
5. Patients must have the following laboratory values as defined in protocol
6. Life expectancy of ≥ 12 weeks
7. Written informed consent obtained

Exclusion Criteria:

1. Patients with evidence of CNS tumor or metastasis
2. Patients with pleural effusion and/or ascites to be drained
3. Patients with any peripheral neuropathy ≥ CTCAE grade 2
4. Impaired cardiac function defined in protocol
5. Acute or chronic liver or renal disease
6. Other concurrent severe and/or uncontrolled medical conditions that could cause unacceptable safety risks or compromise compliance with the protocol
7. Patients who are currently receiving treatment with any of the medications which have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication
8. Patients who have received chemotherapy ≤4 weeks prior to starting study drug or who have not recovered from side effects of such therapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2008-07; Primary Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
To characterize the safety and tolerability of LBH589, including acute and chronic toxicities in Japanese patients with advanced solid tumors. | First cycle

SECONDARY OUTCOMES:
To characterize the pharmacokinetics (PK) of LBH589 | First cycle
To evaluate any antitumor activity of LBH589 in patients with advanced solid tumors | Every 2 cycle

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmeceuticals
Locations (3):
- Japan (3):
  - Novartis Investigational Site, Aichi Prefecture
  - Novartis Investigational Site, Hokkaido
  - Novartis Investigational Site, Hyogo Prefecture

REFERENCES:
- [Derived] Morita S, Oizumi S, Minami H, Kitagawa K, Komatsu Y, Fujiwara Y, Inada M, Yuki S, Kiyota N, Mitsuma A, Sawaki M, Tanii H, Kimura J, Ando Y. Phase I dose-escalating study of panobinostat (LBH589) administered intravenously to Japanese patients with advanced solid tumors. Invest New Drugs. 2012 Oct;30(5):1950-7. doi: 10.1007/s10637-011-9751-0. Epub 2011 Oct 1. PMID 21964801
- See also: Results for CLBH589A1101 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=4467